CLINICAL TRIAL: NCT03894033
Title: Post-market Registry of the AMDS for the Treatment of Acute DeBakey Type I Dissection: PROTECT Registry
Brief Title: Post-market Registry of the AMDS for the Treatment of Acute DeBakey Type I Dissection
Acronym: PROTECT
Status: Active, not recruiting | Type: Observational
Sponsor: JOTEC GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTECT Registry
Record Dates: First submitted 2019-03-27; First posted 2019-03-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Aortic Dissection; Acute DeBakey I Dissection; Acute Type A Dissection; Intramural Hematoma
Keywords: Aortic diseases; Cardiovascular diseases; Aortic Dissection; Aortic Remodeling; Malperfusion; Acute Aortic Dissection
MeSH Terms: conditions — Aortic Dissection; Aortic Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ascyrus Medical Dissection Stent (AMDS) — The device will be implanted during already planned surgical intervention for aortic dissection repair. The participant will be observed and data gathered during the surgery and routine standard of care follow up visits.
  Other Names: AMDS Arch Remodeling Therapy

SUMMARY:
The objective of this registry is to collect information on the performance and clinical benefits of the AMDS (Ascyrus Medical Dissection Stent) to treat patients with acute "DeBakey type I dissections" and with or without so called "preoperative clinically relevant malperfusion" and/or "intramural hematomas".

In a healthy aorta (the vessel that supplies blood to most of the body) the blood flows freely through the main lumen (a space inside the vessel where blood flows). The participants involved in this study have a tear that has separated the inner layer of the aorta wall and created a secondary channel (false lumen) in addition to the main channel (true lumen), and huts, the blood flows through both channels.

AMDS is a stent (a metal tube helping to keep the vessel open) that is placed in the descending thoracic aorta. AMDS is a medical device commercially available in the countries in which the study is being conducted and it is used as standard of care according to its indication.

DETAILED DESCRIPTION:
Observational, prospective and retrospective, non-randomized, non-interventional study to investigate the performance and clinical benefits of the AMDS to treat patients with acute DeBakey type I dissections with or without clinically relevant preoperative malperfusion and/or intramural hematomas (IMH).

Participating physicians will be asked to provide their observations collected during routine care for patients they had decided to treat with AMDS. Informed consent of the patients to allow the use of their clinical records for the purpose of this observational study will be obtained before data are being collected.

A total number of 300 subjects will be enrolled in up to 30 sites in Europe and Canada. The AMDS will be implanted according to the instructions for use and at the discretion of the treating physician.

This registry was initiated by Ascyrus Medical GmbH in August 2019 (DARTS PM Registry). About 70 patients were enrolled at that time by German and Canadian sites under previous protocol. The patient's enrollment was put on-hold and the study has been re-started as PROTECT Registry with updated study documents as per JOTEC's standard operating procedures upon Ethics Committees approvals.

Patients already included in DARTS PM Registry will be re-consented (where applicable as per local regulatory requirements) to allow the retrospective and prospective collection of additional data points not included in the initial version of the protocol. It is also planned to retrospectively include up to 150 subjects of the 300 targeted subjects, which have been treated with AMDS and who consent to the collection of their data (if required by national law) and are willing to continue in this registry, if applicable.

ELIGIBILITY:
Inclusion Criteria

* ≥18 and ≤ 80 years of age (male or female)
* One of the following diagnosed within 14 days:

  * Acute DeBakey type I dissection based on CT angiography; or
  * IMH based on CT angiography

Exclusion Criteria

General Exclusion Criteria:

* < 18 years of age or > 80 years of age (male or female)
* Unwilling to comply with the follow-up schedule
* Refusal to give Informed Consent

Medical Exclusion Criteria:

* Uncontrolled systemic infection
* Uncontrollable anaphylaxis to iodinated contrast
* Known allergy(ies) to nitinol and/ or PTFE
* Patient in extreme hemodynamic compromise requiring cardiopulmonary resuscitation (CPR)
* Preoperative coma

Anatomical Exclusion Criteria:

* Any pathology of mycotic origin
* Subacute or chronic dissection of the ascending aorta and aortic arch (>14 days after the index event)
* Aortic fistulous communication with non-vascular structure (e.g. esophagus, bronchial)
* Extensive thrombus or calcification in the aortic arch as defined by CT angiography
* Excessive tortuosity precluding safe passage of the AMDS as defined by CT angiography

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with Acute DeBakey type I dissection based on CT angiography or IMH based on CT angiography and treated with the AMDS.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Positive arch remodeling | 3-6 months
  Rate of patients with positive arch remodeling defined as either stable or decreasing total aortic diameter in zone 2.

SECONDARY OUTCOMES:
All-cause mortality | In-hospital, at 30 days, 3-6 months, 1 year, 2, 3, 4, 5 years
  Rate of all-cause mortality
Device-related in-hospital mortality | Discharge (definition: between 1-29 days)
  Rate of device-related in-hospital mortality
Device-related mortality | 30 days, 3-6 months, 1 year, 2, 3, 4, 5 years
  Rate of device-related mortality
Resolution of malperfusion in patients who presented initially with malperfusion | Discharge (definition: between 1-29 days), 30 days, and 3-6 months
  Rate of patients with resolution of malperfusion in patients who presented initially with malperfusion
New disabling (Modified Rankin Scale mRS ≥ 2), permanent (>30 days) stroke | Discharge (definition: between 1-29 days), 30 days, 3-6 months,1 year, 2, 3, 4 and 5 years
  Rate of patients with new disabling (mRS ≥ 2), permanent (>30 days) stroke
New disabling (Modified Rankin Scale mRS ≥ 2), transient (< 30 days) stroke | Discharge (definition: between 1-29 days), 30 days, 3-6 months,1 year, 2, 3, 4 and 5 years
  Rate of patients with new disabling (mRS ≥ 2), transient (< 30 days) stroke
New paralysis | Discharge (definition: between 1-29 days), 30 days, 3-6 months,1 year, 2, 3, 4 and 5 years
  Rate of patients with new paralysis
New paraplegia | Discharge (definition: between 1-29 days), 30 days, 3-6 months, 1 year, 2, 3, 4 and 5 years
  Rate of patients with new paraplegia and 5 years
New aortic rupture associated with the implantation of the device | 30 days, 3-6 months,1 year, 2, 3, 4 and 5 years
  Rate of patients with new aortic rupture associated with the implantation of the device (procedure or AMDS related)
Patent innominate artery | Discharge (definition: between 1-29 days), 3-6 months,1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with patent innominate artery (< 50% stenosis of the origin of the branch vessels)
Source of innominate artery stenosis | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Source of innominate artery stenosis (thrombosis, dissection flap covering, dissection extension into vessel)
Patent left carotid artery | Discharge (definition: between 1-29 days), 3-6 months,1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with patent left carotid artery (< 50% stenosis of the origin of the branch vessels)
Source of left carotid artery stenosis | Discharge (definition: between 1-29 days), 3-6 months,1 year, 2, 3, 4 and 5 years (CoreLab)
  Source of left carotid artery stenosis (thrombosis, dissection flap covering, dissection extension into vessel)
Patent left subclavian artery | Discharge (definition: between 1-29 days), 3-6 months,1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with patent left subclavian artery (< 50% stenosis of the origin of the branch vessels)
Source of left subclavian artery stenosis | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Source of left subclavian artery stenosis (thrombosis, dissection flap covering, dissection extension into vessel)
Absence of distal anastomotic new entry tear (DANE) | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4, and 5 years (CoreLab)
  Rate of patients with absence of distal anastomotic new entry tear (DANE)
Increasing true lumen | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4, and 5 years (CoreLab)
  Rate of patients with increasing true lumen [change in diameter at the maximal diameter location within each Zone which is greater than or equal to a 5 mm expansion in comparison to the diameter on the pre-op computed tomography angiography (CTA) scan] in the stented region (Zones 1-3)
Stable true lumen | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4, and 5 years (CoreLab)
  Rate of patients with stable true lumen [change in diameter at the maximal diameter location within each Zone which is between a 5 mm reduction and a 5 mm expansion in comparison to the diameter on the pre-op computed tomography angiography (CTA) scan] in the stented region (Zones 1-3)
Stable or increasing true lumen in the stented region | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with stable or increasing true lumen in the stented region (Zones 1-3)
Decreasing true lumen | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with decreasing true lumen [change in diameter at the maximal diameter location within each Zone which is greater than or equal to a 5 mm reduction in comparison to the diameter on the pre-op computed tomography angiography (CTA) scan] in the stented region (Zones 1-3)
Increasing false lumen | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with increasing false lumen (≥ 5mm) in the stented region (Zones 1-3)
Stable false lumen in the stented region | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with stable false lumen in the stented region (Zones 1-3)
Decreasing false lumen | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with decreasing false lumen (≤ - 5 mm) in the stented region (Zones 1-3)
Rate of patients with stable or decreasing false lumen | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Stable or decreasing false lumen in the stented region (Zones 1-3)
Freedom from AMDS stent removal | Discharge (definition: between 1-29 days), 30 days, 3-6 months, 1 year, 2, 3, 4 and 5 years
  Rate of patients with freedom from AMDS stent removal
Freedom from AMDS-related reintervention | Discharge (definition: between 1-29 days), 30 days, 3-6 months, 1 year, 2, 3, 4 and 5 years
  Rate of patients with freedom from AMDS-related reintervention
Freedom from aortic arch reintervention | Discharge (definition: between 1-29 days), 30 days, 3-6 months, 1 year, 2, 3, 4 and 5 years
  Rate of patients with freedom from aortic arch reintervention
Successful AMDS deployment (at discharge | Discharge (definition: between 1-29 days)
  Rate of patients with successful AMDS deployment (at discharge
Completely thrombosed, partially thrombosed, or patent false lumen in the arch and descending aorta (Zones 0-5) | Discharge (definition: between 1-29 days), 3-6 months, 1 year, 2, 3, 4 and 5 years (CoreLab)
  Rate of patients with completely thrombosed, partially thrombosed, or patent false lumen in the arch and descending aorta (Zones 0-5)

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Kempfert, Prof., Principal Investigator — Deutsches Herzzentrum der Charité
Locations (1):
- Deutsches Herzzentrum der Charité, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
All study participant data will be de-identified.